CLINICAL TRIAL: NCT07229274
Title: Combined Effects of Mulligan Mobilization With Movement and Kinetic Medial Rotation Control for Shoulder on Pain, Range of Motion, and Function Among Fast Bowlers
Brief Title: Effect of Joint Mobilization and Movement Control Exercises on Shoulder Pain and Function in Fast Bowlers (RCT)
Acronym: RCT
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Lahore University of Biological and Applied Sciences (Other)
Responsible Party: Principal Investigator, Hammad Haider, Dr. Hammad Haider, Lahore University of Biological and Applied Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UBAS/ERB/FoRS/25/022
Record Dates: First submitted 2025-10-02; First posted 2025-11-14 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Glenohumeral Internal Rotation Deficit (GIRD)
Keywords: Overhead Athletes; Internal Rotation; Kinetic Control; Sports Injury; Musculoskeletal Disorder
MeSH Terms: conditions — Athletic Injuries; Musculoskeletal Diseases | interventions — Movement

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Movement control exercises with the concept of kinetic control and mobilization with movement (Experimental): Each person will follow this program three times a week. The session starts with a shoulder movement test to check how well the shoulder rotates-60 degrees inward and 45 degrees outward-without the shoulder blade or upper arm moving incorrectly.
  Next, movement retraining exercises are used to fix any incorrect shoulder movements. This includes helping the shoulder and shoulder blade move properly using hands-on support, along with exercises that may be supported or unsupported. Visual cues (like mirrors), touch, and manual guidance are used to teach correct movement.
  Lastly, Mobilization with Movement (MWM) is performed. This involves gently pushing the shoulder joint backward
  Interventions: Other: Kinetic control for shoulder internal rotation with mobilization with movement
- Stretches, strengthening and mobilization with movement (Active Comparator): Each person in the control group will do these exercises three times a week. The session starts with shoulder warm-up exercises like arm circles, shoulder rolls, and reaching overhead. These are done in 2 sets of 10 reps.
  Next is the modified sleeper stretch. This is repeated 3 times, with a 30-second rest between each stretch.
  Then, isometric shoulder exercises are done in standing. The person pushes their arm inward against resistance without actually moving it.
  Finally, Mobilization with Movement (MWM) is used.
  Interventions: Other: stretches, strengthening and mobilization with movement

INTERVENTIONS:
Other: Kinetic control for shoulder internal rotation with mobilization with movement — stretches and strengthening along with mobilization with movement is given to participants. stretches include sleeper stretch and isometrics in strengthening
  Arms: Movement control exercises with the concept of kinetic control and mobilization with movement
Other: stretches, strengthening and mobilization with movement — Each person in the control group will do these exercises three times a week. The session starts with shoulder warm-up exercises like arm circles, shoulder rolls, and reaching overhead. These are done in 2 sets of 10 reps. Next is the modified sleeper stretch. This is repeated 3 times, with a 30-second rest between each stretch. Then, isometric shoulder exercises are done in standing. The person pushes their arm inward against resistance without actually moving it. Finally, Mobilization with Movement (MWM) is used.
  Arms: Stretches, strengthening and mobilization with movement

SUMMARY:
The goal of this clinical trial is to determine combined effects of the Kinetic control for shoulder on pain, range, and function among fast bowlers. The main question it aims to answer is:

Does mulligan mobilization with movement along with kinetic medial rotation control work in decreasing pain, improving shoulder internal range of motion and shoulder function in fast bowlers with glenohumeral internal rotation deficit? Is the combination of Mulligan mobilization with movement along with kinetic control therapy effective in fast bowlers with glenohumeral internal rotation deficit? Treatment arm will receive movement retraining exercises to develop kinetic control with mulligan mobilization and comparison arm will receive standard physical therapy exercises with mulligan mobilization.

Treatment group will receive shoulder warm up exercises, movement retraining exercises and mulligan mobilization with movement.

Comparison group will receive shoulder warm up exercises, modified sleeper stretch, shoulder isometrics and mulligan mobilization with movement.

ELIGIBILITY:
Inclusion Criteria:

* Male cricketers aged 18-45 years.
* Participants experiencing persistent mild to moderate shoulder pain during overhead movements for more than 3 months.
* Fast bowlers actively participating in regular cricket training sessions.
* Presence of Glenohumeral Internal Rotation Deficit (GIRD) greater than 10 degrees, measured with a goniometer by comparing internal rotation of the dominant and non-dominant shoulders.

Exclusion Criteria

* Cricketers who have undergone shoulder (e.g., rotator cuff repair, arthroscopic labrum repair) or elbow surgery within the past 3 months.
* Participants presenting with numbness or tingling sensations in the upper extremity.
* Individuals with comorbidities such as a history of cardiac or pulmonary diseases.
* Subjects with a history of recurrent shoulder dislocations or shoulder instability.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 42 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2026-01-15 (Estimated); Study Completion 2026-02-25 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | baseline, 3 weeks and 6 weeks
  Pain intensity will be evaluated using the Numeric Pain Rating Scale (NPRS) ranging from 0 to 10, where 0 indicates no pain, 1-3 represents mild pain, 4-6 indicates moderate pain, and 7-10 reflects severe pain.
Shoulder Range of Motion | All outcomes will be recorded at baseline, after 3 weeks, and after 6 weeks of intervention.
  Shoulder range of motion will be measured in all planes of movement using a universal goniometer. The movements will include:
  Flexion (0-180°) Extension (0-60°) Abduction (0-180°) Adduction (0-40°) Internal Rotation (0-70°) External Rotation (0-90°) All measurements will be recorded in degrees to assess improvement in joint mobility across these planes.
Functional disability | All outcomes will be recorded at baseline, after 3 weeks, and after 6 weeks of intervention.
  Functional disability will be assessed using the Shoulder Pain and Disability Index (SPADI), which provides a percentage score ranging from 0 to 100%. A low score (0-29%) represents minimal disability, a moderate score (30-59%) indicates moderate disability, and a high score (60-100%) signifies severe functional limitation.

CONTACTS AND LOCATIONS:
Overall Officials: Hammad Haider, MS-MSK PT, Principal Investigator — Lahore University of Biological and Applied Sciences
Locations (2):
- Pakistan (2):
  - Sehat Medical Complex, Lahore, Punjab Province
  - Bata Sports Club, Lahore, Punjab Province

IPD SHARING:
Plan to Share IPD: Undecided